CLINICAL TRIAL: NCT02499640
Title: The Effects of Cold Water Immersion With Different Dosages (Duration and Temperature Variations) on Heart Rate Variability Post-exercise Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paulista University (Other)
Responsible Party: Principal Investigator, Franciele Marques Vanderle, PhD, Paulista University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 51903/2012
Record Dates: First submitted 2015-07-14; First posted 2015-07-16 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Cryotherapy Effect
Keywords: Recovery of function; Autonomic nervous system; Heart rate variability; Cryotherapy; Immersion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- GC (No Intervention): Control group - CG (n = 20), which suffered no recuperative technique
- G1 (Experimental): G1 (n = 20) was subjected to a recovery procedure by immersion cold water for 5 minutes as from 9±1 degrees Celsius
  Interventions: Other: immersion cold water
- G2 (Experimental): G2 (n = 20) was subjected to a recovery procedure by immersion cold water for 5 minutes as from 14±1 degrees Celsius
  Interventions: Other: immersion cold water
- G3 (Experimental): G3 (n = 20) was subjected to a recovery procedure by immersion cold water for 15 minutes as from 9±1 degrees Celsius
  Interventions: Other: immersion cold water
- G4 (Experimental): G4 (n = 20) was subjected to a recovery procedure by immersion cold water for 15 minutes as from 14±1 degrees Celsius
  Interventions: Other: immersion cold water

INTERVENTIONS:
Other: immersion cold water — immersion cold water at different temperatures and exposure times
  Arms: G1; G2; G3; G4

SUMMARY:
The aim of the present study was to investigate the effects of cold water immersion (CWI) during post-exercise recovery with different durations and temperatures on heart rate variability (HRV) indices. 100 participants performed a protocol of jumps and a Wingate test, and immediately afterwards were immersed in cold water, according to the characteristics of each group (CG: control; G1: 5' at 9±1°C; G2: 5' at 14±1°C; G3: 15' at 9±1°C; G4: 15' at 14±1°C). Analyses were performed at baseline, during the recuperative technique (TRec) by CWI and 20, 30, 40, 50 and 60 minutes post-exercise. The HRV indices average of all RR intervals in each analysis period (Mean RR), standard deviation of normal R-R intervals (SDNN), square root of the mean of the sum of the squares of differences between adjacent R-R intervals (RMSSD), spectral components of very low frequency (VLF), low frequency (LF) and high frequency (HF), scatter of points perpendicular to the line of identity of the Poincaré Plot (SD1) and scatter points along the line of identity (SD2) were assessed. Comparisons between groups and moments were performed using the technique of analysis of variance for repeated measures in two scheme factors. A significance level of p<0.05 was considered.

ELIGIBILITY:
Inclusion Criteria:

* male sex
* healthy
* aged between 18 and 30 years
* classified as physically active through the International Physical Activity Questionnaire

Exclusion Criteria:

* smokers
* alcoholics
* use drugs that influenced cardiac autonomic activity
* cardiovascular, metabolic or endocrine diseases.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2014-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in indices of heart rate variability at 60 minutes | 20, 30, 40, 50 and 60 minutes post-exercise